CLINICAL TRIAL: NCT05640726
Title: The First-line Treatment of RCLM With RAS Mutation Was Local Short-course Radiotherapy (SCRT) + PD-1+ Standard Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCO002
Record Dates: First submitted 2022-11-25; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (SCRT) followed by PD-1+ standard therapy (Experimental)
  Interventions: Drug: PD-1; Radiation: SCRT; Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Calcium folinate; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: PD-1 — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks
Radiation: SCRT — Radiotherapy dose: 5×5 Gy
Drug: Bevacizumab — Participants will receive bevacizumab，5mg/kg，intravenously over 60 - 90 minutes, day 1 of every 2 weeks
Drug: Oxaliplatin — Participants will receive Oxaliplatin，85mg/m2，day1
Drug: Calcium folinate — Participants will receive calcium folinate ，400mg/m2，day1
Drug: 5-fluorouracil — Participants will receive 5-fluorouracil ，400mg/m2，day1

SUMMARY:
To explore the efficacy and safety of radiotherapy followed by PD-1+ standard chemotherapy in the first-line treatment of initial unresectable rectal cancer liver metastases

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum；
* The clinical stage evaluated by MRI was T3-4 and/or N+ and M1a(only liver metastasis)；
* ECOG PS 0-2；
* CHild Pugh A；
* Estimated survival ≥3 months;
* Women of childbearing age should comply with contraceptive measures if pregnancy test is negative;
* Adequate organ and bone marrow functions, ecg, blood, biochemical and other basic tests are not contraindications of chemotherapy;
* Adherence to scheduled visits, treatment plans, laboratory tests, and other study procedures Willingness and ability.

Exclusion Criteria:

* Pregnant or lactating women;
* No previous antitumor therapy；
* No previous liver local therapy；
* No contraception during the reproductive period;
* patients known to have a history of allergy to any study drug, similar drug or excipient;
* Patients with risk of massive gastrointestinal bleeding or gastrointestinal obstruction;
* Patients with a history of thromboembolism, except those caused by PICC;
* Patients with active infection;
* Other conditions that the investigator determines are not suitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to 36 months
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival).

SECONDARY OUTCOMES:
objective response rate | every 3 months (up to 36 months）
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate).

IPD SHARING:
Plan to Share IPD: No